CLINICAL TRIAL: NCT03865030
Title: Audiovestibular Manifestations in Patients With Psoriasis
Brief Title: The Inner Ear Function in Psoriatic Patients
Acronym: MP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Paker Miki, principal investigator, Dr. Miki Paker, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0019-19
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: the participants are divided into 2 groups: psoriatic patients and healthy volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- psoriatic patients (Active Comparator): psoriatic patients that are recruited from the dermatology clinic. This arm will undergo audiovestibular evaluation.
  Interventions: Device: audiovestibular function
- healthy volunteers (Active Comparator): Healthy volunteers that are members of the hospital staff and will be recruited from the hospital. This arm will undergo audiovestibular evaluation.
  Interventions: Device: audiovestibular function

INTERVENTIONS:
Device: audiovestibular function — Hearing test- includes a pure tone audiometry, speech audiometry and discrimination level.
  tympanometry- Includes inserting headphones into the participants ears and computer calculation the compliance of the eardrum.
  otoacoustic emission: Includes headphones insertion and calculation of the inner ear audiological function.
  Video head impulse test.
  - Dizziness handicap inventory questionnaire. questionnaire filled by the participants provides a subjective data regarding the severity of the dizziness.

SUMMARY:
Psoriasis in a systemic disease that effects many systems of the body. few studies examined the hearing function of these patients but the results were inconclusive. No study, however, investigated the vestibular function of psoriatic patients.

In a prospective study, the investigators will compare audiovestibular function between psoriatic patients and healthy volunteers. .

DETAILED DESCRIPTION:
Whether psoriatic patients have higher risk for developing inner ear dysfunction (hearing loss and dizziness) is an important issue that needs to be elucidated. Awareness to the elevated risk (if there is any) of inner ear impairment, early detection and treatment of the condition may reduce the morbidities resulting from undiagnosed audiovestibular impairment.

In a prospective study the investigators will examine the inner ear function (vestibular and auditory) of psoriatic patients and compare it to an healthy, young control group.

The study will include 2 groups of participants: psoriatic patients and healthy volunteers. psoriatic patients are recruited from the dermatology clinic while the healthy volunteers are members of the hospital staff.

The participants will undergo 2 sets of examinations:

1. auditory function examination: hearing test (that includes pure tone audiometry, speech audiometry and discrimination level), tympanometry and otoacoustic emissions.
2. vestibular function examination:

   * Video head impulse test: a ten-minute, non- invasive test that includes a computer and a set of goggles worn by the participant. The participants is sitting in front of a wall while wearing the goggles, the investigator moves the participant's head sideways with short, rapid movements. the computer calculates the accuracy and the velocity of the eyes movements.
   * The participants fills a dizziness handicap inventory questionnaire. The participants from the psoriatic group are recruited from the dermatology clinic. The healthy group participants are members of the hospital staff and are recruited from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic patients that are treated in our institute.

Exclusion Criteria:

* Patients suffering from cardiovascular diseases (peripheral vascular disease,congestive heart failure, status post cerebrovascular accident).
* Conditions that are harmful to the inner ear (chronic renal failure,history of noise exposure, usage of ototoxic drugs, chronic otitis media, ear surgery in the past, significant head trauma in the past, ear drum perforation).
* participant that complains of vertigo/ dizziness/ unsteadiness.
* Participant who is/ was suffering from known inner ear disease: meniere disease, acoustic neurinoma, vestibular neuronitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Hearing test | up to 2 weeks after recruitment. estimation time of the outcome is 10 minutes.
  Determining the threshold of each measured tone in decibel units.
Hearing test | up to 2 weeks after recruitment. estimation time of the outcome is 10 minutes.
  Determining the speech threshold in decibel units.
Tympanometry | up to 2 weeks after recruitment. estimation time of the outcome is 3 minutes.
  Determining the type of tympanometry ( one out of the 3 possible options:A,B,C)
Otoacoustic emission | up to 2 weeks after recruitment. estimation time of the outcome is 3 minutes.
  Determining existence or abscence of physiologic otoacoustic emissions in 500, 1000, 2000 Herts.
Video head impulse test | up to 2 weeks after recruitment. estimation time of the outcome is 10 minutes.
  Measuring the velocity of eye movement compared to velocity of the head while the head is thrusted. The measured units are degrees/ seconds
Dizziness handicap inventory | up to 2 weeks after recruitment. estimation time of the outcome is 5 minutes.
  A questionnaire filled out by the participant, assesses subjectively the level of dizziness from which the patient suffers. Score varies between 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Miki Paker, MD, Principal Investigator — haemek medical center
Locations (1):
- Hemek Medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be collected in the principal investigator computer for a period of 7 years.
  The computer has a personal password and the computer if located inside a locked room.

REFERENCES:
- [Background] Pariser DM, Bagel J, Gelfand JM, Korman NJ, Ritchlin CT, Strober BE, Van Voorhees AS, Young M, Rittenberg S, Lebwohl MG, Horn EJ; National Psoriasis Foundation. National Psoriasis Foundation clinical consensus on disease severity. Arch Dermatol. 2007 Feb;143(2):239-42. doi: 10.1001/archderm.143.2.239. PMID 17310004
- [Background] Halligan CS, Bauch CD, Brey RH, Achenbach SJ, Bamlet WR, McDonald TJ, Matteson EL. Hearing loss in rheumatoid arthritis. Laryngoscope. 2006 Nov;116(11):2044-9. doi: 10.1097/01.mlg.0000241365.54017.32. PMID 17075400
- [Background] Bayazit YA, Yilmaz M, Gunduz B, Altinyay S, Kemaloglu YK, Onder M, Gurer MA. Distortion product otoacoustic emission findings in Behcet's disease and rheumatoid arthritis. ORL J Otorhinolaryngol Relat Spec. 2007;69(4):233-8. doi: 10.1159/000101544. Epub 2007 Apr 4. PMID 17409782
- [Background] Dagli M, Sivas Acar F, Karabulut H, Eryilmaz A, Erkol Inal E. Evaluation of hearing and cochlear function by DPOAE and audiometric tests in patients with ankylosing spondilitis. Rheumatol Int. 2007 Apr;27(6):511-6. doi: 10.1007/s00296-006-0249-6. Epub 2006 Nov 9. PMID 17094003
- [Background] Yen YC, Lin YS, Weng SF, Lai FJ. Risk of sudden sensorineural hearing loss in patients with psoriasis: a retrospective cohort study. Am J Clin Dermatol. 2015 Jun;16(3):213-20. doi: 10.1007/s40257-015-0117-9. PMID 25687690
- [Background] Vir D, Sharma P, Mahajan R, Dogra S, Bakshi J, Panda NK. Investigation of high-frequency hearing loss and outer hair cell function of the cochlea in patients with psoriasis: a case-control study. Clin Exp Dermatol. 2019 Jul;44(5):520-523. doi: 10.1111/ced.13805. Epub 2018 Oct 2. PMID 30280411